CLINICAL TRIAL: NCT01226836
Title: Pulmonary Rehabilitation in COPD: the Development and Feasibility of an Education Package
Brief Title: Pulmonary Rehabilitation in Chronic Obstructive Pulmonary Disease (COPD): the Development and Feasibility of an Education Package
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); Belfast Health and Social Care Trust (Other); South Eastern Health and Social Care Trust (Other); Western Health and Social Care Trust (Other)
Responsible Party: Principal Investigator, Brenda O'Neill, Senior Lecturer, Physiotherapy, University of Ulster
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09/0152
Record Dates: First submitted 2010-10-21; First posted 2010-10-22 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Pulmonary Rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Living Well with COPD for Pulmonary Rehabilitation (Experimental)
  Interventions: Other: LWWCOPD for Pulmonary Rehabilitation

INTERVENTIONS:
Other: LWWCOPD for Pulmonary Rehabilitation — As part of clinical care participants will attend a 6 week pulmonary rehabilitation programme consisting of supervised exercise and education sessions. The exercise component will be consistent with the usual pulmonary rehabilitation programme delivered at that site (BTS 2001, NICE 2004). The education sessions will be delivered using the revised LWWCOPD programme (1/week, approx. 30-45min). All health professionals will be provided with the health professionals' manual and supplementary posters for their respective education session. All participants will be provided with the revised LWWCOPD information booklet and an action plan for recognising and managing exacerbations.
  Other Names: LWWCOPD

SUMMARY:
The purpose of this study is to assess the feasibility and acceptability of the revised Living Well With COPD programme (LWWCOPD for Pulmonary Rehabilitation) when used to deliver the education component of pulmonary rehabilitation.

DETAILED DESCRIPTION:
There is limited guidance on what should be included in the education component of pulmonary rehabilitation. International guidelines for COPD and pulmonary rehabilitation suggest numerous topics but do not provide specific information relating to the principal topics and how these should be delivered (BTS 2001, NICE 2004, ATS/ERS 2006). Recently this research team conducted focus groups of patients with COPD and established from their perspective the important education topics that should be covered in pulmonary rehabilitation, along with information on how these should be delivered (Wilson, O'Neill et al. 2008).

The Living Well with COPD (LWWCOPD) programme mostly includes these topics (Bourbeau, Julien et al. 2003). LWWCOPD, which is based on Bandura's self-efficacy theory, has been shown to significantly reduce healthcare utilisation and improve quality of life (Bourbeau, Julien et al. 2003, Bandura 1986). With modification and reformatting, the LWWCOPD programme could be delivered within the structure of pulmonary rehabilitation.

Although the LWWCOPD programme has been previously validated, it is important that the revised version is assessed for feasibility within the context of pulmonary rehabilitation. The practicality of delivering the programme and its acceptance by healthcare providers and patients should be assessed. Therefore, this study will involve a process evaluation to assess the feasibility and acceptability of using the revised LWWCOPD programme (LWWCOPD for Pulmonary Rehabilitation) to deliver the education component of pulmonary rehabilitation in Northern Ireland.

ELIGIBILITY:
Inclusion Criteria:

Participants

* Clinical diagnosis of COPD.
* Good understanding of written English in order to be able to provide accurate feedback on the patient information booklet and material used to facilitate the education sessions (as reported by the individual patient).
* Eligible for pulmonary rehabilitation Health Professionals
* Involved in the delivery of education sessions during pulmonary rehabilitation

Exclusion Criteria:

Participants

* Unable to safely partake in pulmonary rehabilitation (e.g. unstable angina, some musculoskeletal conditions).
* Unable to comprehend or follow instructions (e.g. dementia).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2010-01; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Understanding your COPD questionaire | 6 weeks
  The "Understanding your COPD" questionnaire will be used to assess knowledge, understanding and self-efficacy (pre- and post- pulmonary rehabilitation) and satisfaction with the education sessions (post- pulmonary rehabilitation only). This questionnaire is a self administered questionnaire which takes approximately 10 minutes to complete. It has been developed and assessed for reliability and responsiveness by our research team (Earley, O'Neill et al. 2008).

SECONDARY OUTCOMES:
The Bristol COPD Knowledge Questionnaire (BCKQ) | 6 weeks
  The Bristol COPD Knowledge Questionnaire (BCKQ) will be used to assess knowledge pre- and post- pulmonary rehabilitation (White, Walker et al. 2006). The BCKQ is self-administered and takes 15 minutes to complete. It has been shown to be valid, reliable and responsive in patients with COPD (White, Walker et al 2006).
Global questions | 6 weeks
  The participants will answer three global questions post- pulmonary rehabilitation to assess their perception of the change in their knowledge levels since before the pulmonary rehabilitation programme. The global questions take 1 minute to complete.
Qualitative data collection (patients' perspective) | 6 weeks
  An evaluation questionnaire will be completed after each education session.
Qualitative data collection (health professional's perspective) | 6 weeks
  An evaluation questionnaire will be completed after each education session.

CONTACTS AND LOCATIONS:
Overall Officials: Brenda O'Neill, PhD, Principal Investigator — University of Ulster
Locations (3):
- United Kingdom (3):
  - Belfast Health and Social Care Trust, Belfast, Co ANtrim
  - Southern Eastern Health and Social Care Trust, Belfast
  - Western Health and Social Care Trust, Londonderry

REFERENCES:
- [Background] Wilson JS, O'Neill B, Reilly J, MacMahon J, Bradley JM. Education in pulmonary rehabilitation: the patient's perspective. Arch Phys Med Rehabil. 2007 Dec;88(12):1704-9. doi: 10.1016/j.apmr.2007.07.040. PMID 18047889
- [Derived] Cosgrove D, Macmahon J, Bourbeau J, Bradley JM, O'Neill B. Facilitating education in pulmonary rehabilitation using the living well with COPD programme for pulmonary rehabilitation: a process evaluation. BMC Pulm Med. 2013 Aug 5;13:50. doi: 10.1186/1471-2466-13-50. PMID 23915179